CLINICAL TRIAL: NCT00708175
Title: A Phase 4, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Effect of Pioglitazone Compared to Placebo on Bone Metabolism in Impaired Fasting Glucose, Postmenopausal Women for One Year of Treatment
Brief Title: Efficacy of Pioglitazone on Bone Metabolism in Postmenopausal Women With Impaired Fasting Glucose.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AD-4833_402; U1111-1115-0660 (Registry Identifier: WHO)
Record Dates: First submitted 2008-06-27; First posted 2008-07-02 (Estimated); Results first posted 2012-02-03 (Estimated); Last update posted 2012-02-03 (Estimated); Status verified 2012-01

CONDITIONS: Bone Metabolism
Keywords: Glucose Metabolism Disorder; Dysmetabolic Syndrome; Type II Diabetes; Diabetes Mellitus; Lipoatrophic; Postmenopausal
MeSH Terms: conditions — Glucose Metabolism Disorders; Diabetes Mellitus, Type 2; Diabetes Mellitus | interventions — Pioglitazone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pioglitazone (Experimental)
  Interventions: Drug: Pioglitazone
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Pioglitazone — Pioglitazone 30 mg, tablets, orally, once daily for 4 weeks, then increased to Pioglitazone 45 mg, tablets, orally, once daily for up to 48 weeks.
  Other Names: ACTOS®
  Arms: Pioglitazone
Drug: Placebo — Pioglitazone placebo-matching tablets, orally, once daily for up to 52 weeks.
  Other Names: ACTOS®
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the effect of pioglitazone on bone metabolism in postmenopausal women with impaired fasting glucose.

DETAILED DESCRIPTION:
The World Health Organization has estimated that 30% of all women aged over 50 years (postmenopausal) have osteoporosis according to a definition of Bone Mineral Density at any site being more than 2.5 standard deviations below the mean for young healthy adult women.

A known risk factor for development of osteoporosis and fracture is diabetes mellitus, with correlations to duration of disease and poor glycemic control.

Pioglitazone is a thiazolidinedione developed by Takeda Pharmaceuticals for the treatment of type 2 diabetes. Preclinical studies to date on the bone effects of thiazolidinediones have not clearly identified a mechanism of bone loss. While there is evidence of increased bone fractures in postmenopausal diabetic females treated with a thiazolidinedione, the mechanism is not known. Initial studies with thiazolidinediones in humans have focused on short term exposure (12 to 14 weeks) and non-diabetic females. These studies have shown acute changes in circulating bone markers and bone density, but have been questioned because they may not represent bone metabolism in states of abnormal glucose metabolism. Impaired glucose tolerance has been identified not only as a risk factor for developing type 2 diabetes, but also at higher risk for known complications of diabetes. Examination of the effect of thiazolidinediones on bone metabolism in IGT patients will provide data in patients with abnormal glucose tolerance, but without the potential confounding effects of oral hypoglycemic medications to treat type 2 diabetes.

The primary objective of this study is to evaluate the effect of pioglitazone on bone mass and metabolism in postmenopausal women with impaired fasting glucose or impaired glucose tolerance. Total participation time in this study is approximately 1 year and six months.

ELIGIBILITY:
Inclusion Criteria:

* Is female and has not experienced menses for at least 5 years.
* Has a Fasting Plasma Glucose level greater than or equal to 100 and less than 126 mg/dL or a 2-hour post-oral glucose tolerance test greater than or equal to 140 and less than or equal to 199 mg/dL at Screening.
* Has a body mass index greater than or equal to 16 and less than or equal to 40 kg/m2 and weighs less than 300 pounds (approximately 136 kilograms).
* Agrees to take daily supplements of Vitamin D (a minimum of 800 IU daily) and calcium (a minimum of 1000 mg daily) during the treatment and wash-out periods.
* Has clinical laboratory evaluations (including clinical chemistry, hematology, and complete urinalysis [fasted for at least 8 hours]) within the reference range for the testing laboratory unless the results are deemed not clinically significant by the investigator or sponsor.
* Is in good health as determined by the physician (ie, via medical history and physical examination) at Screening.

Exclusion Criteria:

* Has a fasting triglyceride level greater than 500 mg/dL.
* Has a hemoglobinopathy causing anemia or interfering with glycosylated hemoglobin assays.
* Has an alanine transaminase level greater than or equal to 2.5 times the upper limit of normal, active liver disease or jaundice.
* Has Vitamin D (25-OH-D) less than 20 ng/mL.
* Has Baseline Bone Mineral Density defined as a T-score less than -2.0 at the total hip, spine, or femoral neck based on Caucasian reference values.
* Has unexplained microscopic or macroscopic hematuria confirmed by repeat testing.
* Has any of the following disorders:

  * Rheumatoid Arthritis
  * Thyroid (uncontrolled on thyroid replacement therapy), parathyroid, pituitary, nutritional, inflammatory, gastrointestinal, autoimmune, or renal or other disease known to affect bone metabolism.
  * A personal history of kidney stones.
* Has a clinical history after age 45 of wrist, hip, or leg fractures.
* Has a history of more than 1 asymptomatic vertebral deformity or any vertebral deformity attributed to osteoporosis.
* Has a known history of drug abuse (defined as illicit drug use) or a known history of alcohol abuse within 2 years of Screening.
* Has signs and/or symptoms of heart failure.
* Is currently participating in another investigational study or has participated in an investigational study within the past 30 days or 5 half lives of the investigational product, whichever is longer.
* Has any other serious disease or condition at screening or at randomization that might make it difficult to successfully manage and follow up with the subject according to the protocol.
* Has a history of cancer, other than basal cell carcinoma or Stage 1 squamous cell carcinoma of the skin that has not been in remission for at least 5 years prior to the first dose of study drug.
* Has a history of breast cancer.
* Is taking or has ever taken pioglitazone or other Thiazolidinediones.
* Has received or donated blood or blood products within 30 days preceding the Screening visit or plans to donate blood during the study.

Max Age: 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 156 (Actual)
Dates: Start 2008-05; Primary Completion 2011-01 (Actual); Study Completion 2011-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: VP Clinical Science Strategy, Study Director — Takeda
Locations (34):
- United States (34):
  - Greenbrae, California
  - Los Banos, California
  - San Diego, California
  - Walnut Creek, California
  - West Hills, California
  - Lakewood, Colorado
  - Longmont, Colorado
  - Boynton Beach, Florida
  - Hialeah, Florida
  - Jupiter, Florida
  - Dunwoody, Georgia
  - Gainesville, Georgia
  - Honolulu, Hawaii
  - Idaho Falls, Idaho
  - Chicago, Illinois
  - Des Moines, Iowa
  - Iowa City, Iowa
  - Louisville, Kentucky
  - Metarie, Louisiana
  - Scarborough, Maine
  - Bethesda, Maryland
  - Detroit, Michigan
  - Omaha, Nebraska
  - Albuquerque, New Mexico
  - Mineola, New York
  - West Haverstraw, New York
  - Pinehurst, North Carolina
  - Cincinnati, Ohio
  - Portland, Oregon
  - Aiken, South Carolina
  - Greenville, South Carolina
  - Brentwood, Tennessee
  - Denton, Texas
  - Houston, Texas

REFERENCES:
- [Derived] Ipsen EO, Madsen KS, Chi Y, Pedersen-Bjergaard U, Richter B, Metzendorf MI, Hemmingsen B. Pioglitazone for prevention or delay of type 2 diabetes mellitus and its associated complications in people at risk for the development of type 2 diabetes mellitus. Cochrane Database Syst Rev. 2020 Nov 19;11(11):CD013516. doi: 10.1002/14651858.CD013516.pub2. PMID 33210751
- [Derived] Bone HG, Lindsay R, McClung MR, Perez AT, Raanan MG, Spanheimer RG. Effects of pioglitazone on bone in postmenopausal women with impaired fasting glucose or impaired glucose tolerance: a randomized, double-blind, placebo-controlled study. J Clin Endocrinol Metab. 2013 Dec;98(12):4691-701. doi: 10.1210/jc.2012-4096. Epub 2013 Sep 20. PMID 24057294
- See also: ACTOS® Package Insert — http://general.takedapharm.com/content/file/pi.pdf?applicationcode=ab2d7112-8eb3-465a-8fda-35018a9eafb0&fileTypeCode=ACTOSPI

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 25 investigative sites in the United States from 23 May 2008 to 02 February 2011.
Pre-assignment Details: Postmenopausal participants enrolled in 1 of 2 treatment groups to examine the effect of pioglitazone on bone mineral density (BMD) by dual-energy-ray absorptiometry (DXA). Participants with >7% decrease from baseline in BMD of the total proximal femur or spine based on DXA scan results (confirmed with a repeat scan) were to discontinue study drug.
Period: Overall Study
Arm/Group | Pioglitazone | Placebo
Started | 78 | 78
Completed | 60 | 57
Not Completed | 18 | 21
Not completed — Adverse Event | 4 | 5
Not completed — Protocol Violation | 2 | 3
Not completed — Lost to Follow-up | 5 | 3
Not completed — Withdrawal by Subject | 5 | 7
Not completed — BMD loss >7% | 2 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pioglitazone | Placebo | Total
Number analyzed (Participants) | 78 | 78 | 156
Age Continuous [Mean (Standard Deviation); unit: years] | 59.0 (5.04) | 60.2 (6.17) | 59.6 (5.65)
Age, Customized [Number; unit: participants]
  <45 years | 0 | 1 | 1
  Between 45 and 64 years | 66 | 54 | 120
  ≥65 years | 12 | 23 | 35
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 78 | 78 | 156
  Male | 0 | 0 | 0
Race (NIH/OMB) [Number; unit: participants] — For race, a participant may choose more than one category for race. Participants who indicated more than one race category are included in each category indicated and they are also included in the Multiracial category. Thus the total number and percentage of participants does not necessarily add up to the total number of randomized participants.
  participants
    American Indian or Alaska Native | 1 | 0 | 1
    Asian | 2 | 4 | 6
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Black or African American | 6 | 6 | 12
    White | 70 | 68 | 138
    More than one race | 1 | 0 | 1
    Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 78 | 78 | 156
Ethnicity [Number; unit: participants]
  Hispanic or Latino | 38 | 34 | 72
  Non Hispanic or Latino | 40 | 44 | 84
Height [Mean (Standard Deviation); unit: cm] | 160.3 (6.85) | 161.1 (7.70) | 160.7 (7.28)
Weight [Mean (Standard Deviation); unit: kg] | 76.03 (13.406) | 79.02 (16.326) | 77.53 (14.964)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m2] | 29.61 (5.055) | 30.29 (4.872) | 29.95 (4.960)
Smoking Classification [Number; unit: participants]
  Never smoked | 52 | 55 | 107
  Current smoker | 7 | 9 | 16
  Ex-smoker | 19 | 14 | 33
History of hip fracture? [Number; unit: participants]
  Yes | 5 | 3 | 8
  No | 73 | 75 | 148

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline to Month 12 in Bone Mineral Density in the Total Proximal Femur by Dual-Energy-Ray Absorptiometry (DXA)
Description: The change in bone mineral density in the total proximal femur at month 12 relative to baseline. DXA is a means of measuring BMD through x-ray.
Time Frame: Baseline and Month 12.
Population: All randomized participants who received at least 1 dose of study medication (Full Analysis Set). This was an observed case analysis with no imputation for missing data. If a valid pre-treatment scan was not available, the earliest (within 30 days) post-dosing scan was used as Baseline. There was one such participant for this endpoint.
Measure: Least Squares Mean (Standard Error); unit: percent
Arm/Group | Pioglitazone | Placebo
Number analyzed (Participants) | 58 | 61
percent | -0.69 (0.284) | -0.14 (0.277)
Statistical Analysis 1: Comparison: Pioglitazone vs Placebo; The sample size was calculated using a precision approach to estimate the difference between the pioglitazone and placebo treatment groups in the percent change from baseline in BMD; Test type: Superiority or Other; p = 0.170, ANCOVA — P-value is from a 1-way ANCOVA with treatment group as a factor and baseline BMD as a covariate. There were no multiplicity adjustments; Mean Difference (Final Values) = -0.55, 95% CI 2-sided [-1.33 to 0.24]

2. Secondary Outcome: Percent Change From Month 12 to Month 18 in Bone Mineral Density in the Total Proximal Femur by DXA
Description: The change in bone mineral density in the total proximal femur at month 18 relative to month 12. DXA is a means of measuring BMD through x-ray.
Time Frame: Month 12 and Month 18.
Population: All randomized participants who received at least 1 dose of study medication (Full Analysis Set). This was an observed case analysis with no imputation for missing data.
Measure: Least Squares Mean (Standard Error); unit: percent
Arm/Group | Pioglitazone | Placebo
Number analyzed (Participants) | 53 | 56
percent | -0.14 (0.265) | 0.04 (0.258)
Statistical Analysis 1: Comparison: Pioglitazone vs Placebo; Test type: Superiority or Other; p = 0.640, ANCOVA — P-value is from a 1-way ANCOVA with treatment group as a factor and the Month 12 BMD value as a covariate. There were no multiplicity adjustments; Mean Difference (Final Values) = -0.17, 95% CI 2-sided [-0.91 to 0.56]

3. Other Pre Specified Outcome: Change in Fasting Plasma Glucose (FPG)
Description: The change between the fasting plasma glucose value collected at each time frame indicated.
Time Frame: Baseline and Month 12; Month 12 and Month 18.
Population: All randomized participants who received at least 1 dose of study medication (Full Analysis Set).
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Pioglitazone | Placebo
Number analyzed (Participants) | 78 | 78
mg/dL
  Baseline to Month 12 (n=57; n=61) | -2.8 (1.66) | 6.0 (1.61)
  Month 12 to Month 18 (n=54; n=57) | 0.4 (2.00) | -1.0 (1.94)

4. Other Pre Specified Outcome: Number of Participants Who Converted to Type 2 Diabetes Mellitus (T2DM)
Description: Participants were considered to have converted to T2DM if there were ≥2 consecutive post-Baseline FPG measurements ≥126 mg/dL. Participants meeting criteria were tabulated and summarized by Study Period (Treatment and Follow-up). Conversion to T2DM during Treatment Period occurred if either both of the consecutive post-Baseline high FPG values, or the first of the 2 consecutive high values occurred on or before the first day off study drug. Conversion to T2DM occurred during the Follow-up Period if both consecutive high values occurred after at least 1 day after the Treatment Period.
Time Frame: Up to 18 months.
Population: All randomized participants who received at least 1 dose of study medication (Full Analysis Set).
Measure: Number; unit: participants
Arm/Group | Pioglitazone | Placebo
Number analyzed (Participants) | 78 | 78
participants
  Double-Blind Period (n=76; n=75) | 1 (1.3) | 7 (9.3)
  Follow-up Period (n=63; n=59) | 0 (0.0) | 1 (1.7)

5. Other Pre Specified Outcome: Number of Participants With Fracture
Description: Number of participants with confirmed (through an adjudication process) fractures during the study. Circumstances surrounding the fracture, available X-ray and other diagnostic results and healing status were collected for the adjudication process.
Time Frame: Up to 18 months.
Population: All randomized participants who received at least 1 dose of study medication (Full Analysis Set).
Measure: Number; unit: participants
Arm/Group | Pioglitazone | Placebo
Number analyzed (Participants) | 78 | 78
participants | 1 | 3

ADVERSE EVENTS:
Time Frame: Treatment-emergent serious adverse events are serious adverse events that started after the first dose of study drug and no more than 30 days after the last dose of study drug.
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | Pioglitazone | Placebo
Serious Adverse Events (participants affected / at risk) | 3/78 | 1/78
Other Adverse Events (participants affected / at risk) | 32/78 | 34/78
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pioglitazone (N=78) | Placebo (N=78)
Cardiac failure congestive (Cardiac disorders) | 1 | 0
Diverticulitis (Infections and infestations) | 1 | 0
Peridiverticular abscess (Infections and infestations) | 1 | 0
Tracheobronchitis (Infections and infestations) | 0 | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 1 | 0
Migraine (Nervous system disorders) | 1 | 0
Calculus urinary (Renal and urinary disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Pioglitazone (N=78) | Placebo (N=78)
Urinary tract infection (Infections and infestations) | 6 | 10
Oedema peripheral (General disorders) | 9 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 | 4
Sinusitis (Infections and infestations) | 0 | 6
Back pain (Musculoskeletal and connective tissue disorders) | 4 | 5
Cough (Respiratory, thoracic and mediastinal disorders) | 5 | 0
Blood glucose increased (Investigations) | 1 | 4
Blood parathyroid hormone increased (Investigations) | 4 | 1
Fall (Injury, poisoning and procedural complications) | 2 | 4
Headache (Nervous system disorders) | 2 | 4
Influenza (Infections and infestations) | 0 | 4
Nausea (Gastrointestinal disorders) | 4 | 2
Weight increased (Investigations) | 4 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.